CLINICAL TRIAL: NCT01889485
Title: Screening and Access to Health Care for Vascular Disease in Urban and Suburban Patient Populations
Brief Title: Screening and Access to Health Care for Vascular Disease
Status: Completed | Type: Observational
Sponsor: Endeavor Health (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: EH12-224
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-06

CONDITIONS: Aortic Aneurysm, Abdominal; Carotid Stenosis; Peripheral Arterial Disease
Keywords: Aortic Aneurysm, Abdominal; Carotid Stenosis; Peripheral Arterial Disease; Health Services Accessibility
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Carotid Stenosis; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a pilot study designed to validate our methods of recruitment, screening and data collection in the community. The project will help to establish the feasibility of the study design to lay the groundwork for a potentially larger study. The final study will allow us to estimate the incidence and prevalence of abdominal aortic aneurysm (AAA), carotid artery stenosis, and peripheral artery disease (PAD) in different geographic areas in a large urban setting, as well as determine patient access to healthcare and treatment for vascular disease as related to geographic and racial differences.

ELIGIBILITY:
Inclusion Criteria:

* age 55 or older
* willing/able to provide consent
* willing to participate in follow-up phone calls at defined intervals for up to 5 years

Exclusion Criteria:

* unable to provide consent to participate
* unwilling/unable to participate in the follow-up phone call

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer subjects age 55 and over who sign informed consent will be enrolled in three separate neighborhoods in the Chicago area (North, South, West).
Sampling Method: Non-Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Geographic and racial differences in access to follow-up care if significant disease is identified through the screening event | 5 years

SECONDARY OUTCOMES:
Geographical and racial differences in patterns of accessing healthcare prior to the screening events. | 1 year
Differences in rates of interventions throughout the 5 year follow-up period. | 5 years
Differences in the rates of complications related to treatment of vascular disease in the various geographic areas in which the events are held. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Omar Morcos, MD, Principal Investigator — Endeavor Health
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

DOCUMENTS (1):
  • Informed Consent Form (2014-04-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT01889485/ICF_000.pdf